CLINICAL TRIAL: NCT01200446
Title: Docosahexaenoic Acid (DHA) as a Nutritional Treatment for Exercise-Induced Bronchoconstriction and Airway Inflammation in Asthma
Brief Title: Effect of a Component of Fish Oil on Exercise-Induced Bronchoconstriction and Airway Inflammation in Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Timothy Mickleborough, PhD / Associate Professor, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1005001346
Record Dates: First submitted 2010-09-01; First posted 2010-09-13 (Estimated); Last update posted 2011-05-26 (Estimated); Status verified 2011-05

CONDITIONS: Asthma
Keywords: Asthma; Exercise-Induced Bronchoconstriction; Inflammation; Airway; Fish Oil; Docosahexaenoic Acid; DHA
MeSH Terms: conditions — Asthma; Inflammation | interventions — Docosahexaenoic Acids; Corn Oil; Soybean Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Docosahexaenoic Acid (DHA) (Placebo Comparator): Eight subjects will take 8 placebo DHA capsules per day for 3 weeks.
  Interventions: Dietary Supplement: Placebo Docosahexaenoic Acid
- Active Docosahexaenoic Acid (DHA) (Experimental): Eight subjects will take 8 active DHA capsules per day for 3 weeks.
  Interventions: Dietary Supplement: Docosahexaenoic Acid

INTERVENTIONS:
Dietary Supplement: Docosahexaenoic Acid — 8 docosahexaenoic acid (4.0 grams) capsules per day for 3 weeks.
  Other Names: DHA
  Arms: Active Docosahexaenoic Acid (DHA)
Dietary Supplement: Placebo Docosahexaenoic Acid — 8 placebo docosahexaenoic acid (corn and soy oil blend) capsules per day for 3 weeks.
  Other Names: Corn Oil; Soy Oil
  Arms: Placebo Docosahexaenoic Acid (DHA)

SUMMARY:
Docosahexaenoic acid (DHA) is a component of fish oil that is known to support a healthy cardiovascular system, maintain brain function, reduce depression, and improve inflammatory diseases. The study hypothesis is that DHA supplementation will diminish exercise-induced bronchoconstriction and airway inflammation as compared to placebo.

DETAILED DESCRIPTION:
To date, fish oil supplementation studies in patients with asthma have used a combination of omega-3 polyunsaturated fatty acids. A study on the specific formula that is most effective in preventing exercise-induced bronchoconstriction (EIB) has yet to be conducted in humans. Nevertheless, it has been shown that a docosahexaenoic acid (DHA) metabolite, protectin D1, is involved in the active resolution of airway inflammation and that its concentration is greater in healthy control subjects' exhaled breath condensates as compared to patients with asthma during a clinical exacerbation. Supplementing asthmatics with DHA could enable an increased availability of protectin D1 to help resolve airway inflammation during an asthma attack. Furthermore, DHA is known to support a healthy cardiovascular system, maintain brain function, and reduce depression in addition to alleviating inflammatory diseases. Thus, pure DHA supplementation could help patients manage their asthma while providing for their overall health.

The main aim of this study is to determine whether pure DHA can attenuate EIB and airway inflammation in adults with asthma. It is hypothesized that DHA supplementation will diminish EIB and airway inflammation compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma, based on medication use as well as history and symptoms as outlined in the NHLBI Guidelines for the Diagnosis and Management of Asthma
* Diagnosis of EIB, based on a ≥10% fall in FEV1, a measure of lung function, after dry air eucapnic voluntary hyperventilation (EVH), a simulated exercise challenge
* Not currently taking asthma maintenance medication or physician approval to discontinue current asthma medication for the duration of the study
* Not currently taking any fish oil supplements above the level recommended for adequate intake (if currently taking supplements, can participate if the subject stops taking the supplements for 2 weeks before starting the study and throughout the study)
* Agree to limit fish consumption to 1 fish meal per week throughout the study

Exclusion Criteria:

* Post-EVH FEV1 (the amount of air blown out in the first second of a forced exhalation) decreases by more than 50% compared to the subject's resting FEV1 at the first lab testing session
* Pregnancy
* History of cardiovascular disease, including hyperlipidemia (high cholesterol) and hypertension (high blood pressure)
* History of bleeding disorders or delayed clotting time
* History of diabetes
* History of seizures
* Allergy to fish oil
* Allergy to corn or soy products (placebo is a mixture of corn and soy oil)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function (Percent Change in FEV1, measured in Liters) | 8 weeks
  The percent change in FEV1 is the percent change in the volume of air exhaled during the first second of a forced exhalation as measured before and after the surrogate exercise challenge.

SECONDARY OUTCOMES:
DHA Metabolite Concentration in Exhaled Breath Condensate | 8 weeks
  The concentration (ng/mL) of the DHA metabolites protectin D1 and 17S-hydroxy-docosahexaenoic acid in exhaled breath condensate will be measured using liquid chromatography.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy D Mickleborough, PhD, Study Director — Indiana University
Locations (1):
- Indiana University, Bloomington, Indiana, United States

REFERENCES:
- [Background] Mickleborough TD, Murray RL, Ionescu AA, Lindley MR. Fish oil supplementation reduces severity of exercise-induced bronchoconstriction in elite athletes. Am J Respir Crit Care Med. 2003 Nov 15;168(10):1181-9. doi: 10.1164/rccm.200303-373OC. Epub 2003 Aug 6. PMID 12904324
- [Background] Mickleborough TD, Lindley MR, Ionescu AA, Fly AD. Protective effect of fish oil supplementation on exercise-induced bronchoconstriction in asthma. Chest. 2006 Jan;129(1):39-49. doi: 10.1378/chest.129.1.39. PMID 16424411